CLINICAL TRIAL: NCT01411553
Title: ECG Leadwires: Do Disposable Leadwires Reduce the Incidence of Bacterial Infections in ICU Patients and Provide Adequate Signaling in Stepdown/Telemetry Environment Compared to Cleaned Reusable ECG Leadwires?
Brief Title: ECG Leadwires: Disposable Versus Cleaned, Reusable
Acronym: ECG-LW
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Nancy M. Albert, Ph.D., Senior Director, Nursing Research and Innovation, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: clevelandCF
Record Dates: First submitted 2011-08-05; First posted 2011-08-08 (Estimated); Last update posted 2016-02-23 (Estimated); Status verified 2016-02

CONDITIONS: Critically Ill Patients; Cardiovascular Surgery Telemetry Patients
Keywords: ICU; Telemetry; ECG lead wire monitoring; Infection; Nuisance alarms
MeSH Terms: conditions — Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Reusable ECG leadwires-ICU (No Intervention): Current ECG leadwires will be used
- Disposable ECG leadwires-ICU (Active Comparator): Disposable ECG-LW
  Interventions: Other: Disposable ECG-LW

INTERVENTIONS:
Other: Disposable ECG-LW — Disposable ECG leadwires used in ICU and telemetry monitoring; 5 lead sets for ICU and 6-lead sets for telemetry
  Other Names: Covidien disposable ECG lead wires
  Arms: Disposable ECG leadwires-ICU

SUMMARY:
Null hypothesis: (1) there is no difference in rates of ICU-acquired infection based on using disposable or cleaned, reusable ECG leadwires and (2) In cardiac surgical telemetry floors, there is no difference in false or nuisance sightings or crisis calls based on using disposable or cleaned, reusable ECG leadwires.

DETAILED DESCRIPTION:
Primary purposes: Using a randomized controlled trial methodology and randomizing similar (matched) intensive care units (ICU) to either disposable or cleaned, reusable ECG-LW: 1. Is there a difference in the rate of blood stream infection (BSI) and ventilator-associated pneumonia (VAP) in ICU environments (medical ICU, surgical ICU, cardiothoracic ICU, and neuroscience ICU) and surgical site infection (SSI); specifically, sternal wound infections in cardiothoracic ICU that utilize disposable vs. cleaned, reusable ECG-LW? 2. Is there a difference in ICU length of stay based on ECG-LW used: disposable vs. cleaned, reusable? 3. After controlling for patient age, comorbidity index and after removing patients who's date of BSI or VAP infections were within 48 hours of admission to the ICU, is there a difference in the rate of (A) blood stream infection (BSI), (B) ventilator-associated pneumonia (VAP) and (C) SSI in ICU environments (when applicable) that utilize disposable vs. cleaned, reusable ECG-LW? Secondary purposes: Using a randomized controlled trial methodology and randomizing similar telemetry units to either disposable or cleaned, reusable ECG-LW: 1. Is there a difference in the number of false/nuisance sightings/crisis calls (i.e., lead off, no telemetry, lead failure or other false alarms) identified by the Central Monitoring Unit (CMU)? 2. Is there a difference in true sightings/crisis calls identified by the CMU based on unit assignment of disposable or cleaned, reusable ECG-LW? 2b. If yes to #2, is there a difference in types of true sightings/calls identified by the CMUbased on assignment of disposable or cleaned, reusable ECG-LW?

ELIGIBILITY:
Inclusion Criteria:

* Primary HO: patients treated in an ICU setting; Secondary HO: Patients treated in cardiac telemetry setting

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 4056 (Actual)
Dates: Start 2011-09; Primary Completion 2012-12 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Blood stream infection | 7 months
  culture findings

SECONDARY OUTCOMES:
false/nuisance alarms | 4 months
  alarms generated by ECG tracings due to various causes (leads off, leads crimped, etc)

CONTACTS AND LOCATIONS:
Overall Officials: Nancy M Albert, PhD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States